CLINICAL TRIAL: NCT06841562
Title: Targeted Remotely-delivered Anti-inflammatory Interventions With Exercise for Rheumatoid Arthritis - Early Rheumatoid Arthritis Pilot Study
Brief Title: Targeted Remotely-delivered Anti-inflammatory Interventions With Exercise for Rheumatoid Arthritis
Acronym: TRAINERa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00117047
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: exercise training
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRAINERa intensive exercise training (Experimental): Participants with early and active rheumatoid arthritis (RA) will complete a 12-week RA-tailored remotely supervised and delivered moderate to vigorous intensity aerobic training combined with resistance training exercise program.
  Interventions: Behavioral: TRAINERa intensive exercise training

INTERVENTIONS:
Behavioral: TRAINERa intensive exercise training — Remotely-delivered exercise training intervention

SUMMARY:
The primary objective of this study is to assess the feasibility of an intensive, remotely-delivered, combined aerobic and resistance training exercise program for patients with Rheumatoid Arthritis (RA) and to collect data to support power calculations for a larger research study.

DETAILED DESCRIPTION:
The primary aim of this study is to assess the feasibility of an intensive, remotely-delivered, combined aerobic and resistance training exercise intervention program for patients with Rheumatoid Arthritis (RA) and to collect data to inform the design of a larger research study. This protocol will build upon a recent project, gathering additional data to support future grant applications. The findings will provide critical information for determining the design and appropriate sample size and ensuring sufficient statistical power for a larger study. Additionally, this pilot will evaluate the practicality of implementing a remotely supervised exercise training intervention in early and active RA patients, helping to establish its potential for broader clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Persons with early RA - defined as duration of diagnosis equal to or less than 6 months, and prior to starting biologic DMARD therapy. Participants may be on one or a combination of the following conventional synthetic DMARDs: hydroxychloroquine, methotrexate, sulfasalazine, leflunomide, azathioprine
* Seropositive (positive rheumatoid factor or anti-citrullinated protein antibody) or erosions typical of RA on radiographs
* History of fulfilling 2010 ACR/EULAR Classification Criteria for RA
* Active RA, not in clinical disease remission (Clinical Disease Activity Index for RA (CDAI) > 2.8)
* Stable doses (for ≥ 1 month) of all RA and cardiovascular risk-related medications (including statins, metformin, SGLT2 inhibitors, GLP1RA) except for glucocorticoids

Exclusion Criteria:

* Pregnant or intending to become pregnant during the intervention period
* Current treatment with exogenous insulin
* Other inflammatory arthropathy or myopathy, Paget's disease, pigmented villonodular synovitis, joint infection, ochronosis, neuropathic arthropathy, osteochondromatosis, acromegaly, hemochromatosis, or Wilson's disease
* Current malignancy other than minimally invasive carcinomas routinely treated topically or with minor surgical treatment
* Absolute contraindications to exercise testing: ongoing unstable angina; uncontrolled cardiac arrhythmia with hemodynamic compromise; active endocarditis; symptomatic severe aortic stenosis; decompensated heart failure; acute pulmonary embolism, pulmonary infarction, or deep vein thrombosis; acute myocarditis or pericarditis; acute aortic dissection; physical disability that precludes safe and adequate testing
* Relative contraindications to exercise testing: known obstructive left main coronary artery stenosis; moderate to severe aortic stenosis with uncertain relation to symptoms; tachyarrhythmias with uncontrolled ventricular rates; acquired advanced or complete heart block; hypertrophic obstructive cardiomyopathy with severe resting gradient; recent stroke or transient ischemic attack; mental impairment with limited ability to cooperate; uncorrected medical conditions, such as hypertension (see below), significant anemia, important electrolyte imbalance, and hyperthyroidism
* Acute myocardial infarction (MI) within six months
* Resting hypertension with systolic or diastolic blood pressures >160/90 mm Hg
* Lack of internet access
* Planned, intentional weight loss during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of exercise training intervention | The primary feasibility target is participant adherence to the intervention protocol exercise prescription averaged over the course of the final 6 weeks of the 12-week program > 60%.
  Feasibility will be measured as a dichotomous outcome through patient adherence, defined as meeting 100% of the prescribed exercise protocol, on average.

SECONDARY OUTCOMES:
Acceptability of exercise training intervention | 12 weeks
  Acceptability will be measured with dichotomous patient-reported responses to questions on willingness to recommend the current intervention to others with RA and willingness to participate in such a study again.
Safety of exercise training intervention | 12 weeks
  Safety will be measured by adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Andonian, MD, MHSc, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
New clinical data will be collected from 15 participants with rheumatoid arthritis before and after a 12-week exercise training intervention. All de-identified individual participant data (including demographic, clinical and immune cell data) will be deposited into a NIH supported public repository. Adequate information will be retained to generate a unique identifier for each study participant.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All scientific data from this project will be made available by the end of the award period or time of associated publication, whichever comes first.

REFERENCES:
- [Background] Andonian BJ, Ross LM, Sudnick AM, Johnson JL, Pieper CF, Belski KB, Counts JD, King AP, Wallis JT, Bennett WC, Gillespie JC, Moertl KM, Richard D, Huebner JL, Connelly MA, Siegler IC, Kraus WE, Bales CW, Porter Starr KN, Huffman KM. Effect of Remotely Supervised Weight Loss and Exercise Training Versus Lifestyle Counseling on Cardiovascular Risk and Clinical Outcomes in Older Adults With Rheumatoid Arthritis: A Randomized Controlled Trial. ACR Open Rheumatol. 2024 Mar;6(3):124-136. doi: 10.1002/acr2.11639. Epub 2023 Dec 21. PMID 38126260